CLINICAL TRIAL: NCT06040840
Title: WALANT Versus Axillary Brachial Plexus Block in Carpal Tunnel Release: a Non-inferiority Randomized Controlled Trial
Brief Title: WALANT Versus Axillary Brachial Plexus Block in Carpal Tunnel Release
Acronym: WALAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2023/02
Record Dates: First submitted 2023-09-07; First posted 2023-09-18 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Carpal Tunnel Syndrome
Keywords: WALANT; Axillary block; Regional anesthesia; Tourniquet; Carpal Tunnel Release; Postoperative analgesia; Perioperative patient satisfaction
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Tourniquets; Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BAX group (Active Comparator): Axillary brachial plexus block + Tourniquet
  Interventions: Procedure: BAX; Procedure: Tourniquet; Drug: Lidocaine
- WALANT group (Experimental): Wide Awake Local Anesthesia No Tourniquet
  Interventions: Procedure: WALANT; Drug: Lidocaine + Epinephrine

INTERVENTIONS:
Procedure: BAX — Injection of 30 mL of lidocaine (10 mg/ml) around the median, radial, ulnar and musculocutaneous nerves.
  Arms: BAX group
Procedure: Tourniquet — Inflation pressure 75 to 100 mmHg above the patient's systolic blood pressure.
  Arms: BAX group
Drug: Lidocaine — Axillary block with Lidocaine (10 mg/ml).
  Arms: BAX group
Procedure: WALANT — Preparation of a mixture of 20 ml of lidocaine (10 mg/ml) with epinephrine (0.005 mg/ml) + 3 ml Na bicarbonate (84 mg/ml) + 17 ml sterile normal saline.
  The ultrasound probe will be placed to obtain a transverse image of the median nerve at the wrist. With an in-plane technique, a 50mm ultrasound needle (Ultraplex 360°, B Braun, Melsungen, Germany) will be advanced to achieve a spread of 5 ml of the solution posterior and then anterior to the median nerve under the annular carpal ligament.
  Then the ultrasound probe will be placed to obtain a longitudinal image of the median nerve at the wrist. With an in-plane technique, a 50mm ultrasound needle (Ultraplex 360°, B Braun, Melsungen, Germany) will be advanced to achieve a spread of 15 ml of the solution anterior to the median nerve towards the carpal tunnel.
  At last, a local infiltration with 5 ml of the solution will be performed around the surgical incision.
  Arms: WALANT group
Drug: Lidocaine + Epinephrine — WALANT technique with lidocaine (10 mg/ml) combined with 0.005 mg/ml epinephrine.
  Arms: WALANT group

SUMMARY:
Carpal tunnel syndrome (CTS) is a common medical condition that remains one of the most frequently reported forms of median nerve compression. Surgical procedure is a treatment option for CTS. For this surgery of the upper extremity, regional anesthesia (RA) is the strategy that should be systematically preferred because it is associated with shorter postanesthetic care and less pain compared to general anesthesia. Multiple approaches to block the brachial plexus are available for the surgery of the upper extremity below the elbow, but the axillary block (BAX) remains the most common approach as it is associated with low side effects.

One of the most significant recent advances in the surgery of the upper extremity has been the emergence of Wide-Awake Local Anesthesia No Tourniquet (WALANT) technique. WALANT is an infiltration technique of a local anesthetic (LA) (lidocaine) and a hemostatic agent (epinephrine) directly into the operative site to induce anesthesia and hemostasis in the area of the surgical procedure to provide conditions suitable for hand surgery without sedation and tourniquet. Given its effectiveness and low side effects, WALANT could be a technique of choice in ambulatory surgery.

The main objective of this non-inferiority, prospective, randomized, open-label, parallel-group controlled trial is to assess the efficacy of WALANT technique compared to BAX in carpal tunnel release (CTR).

DETAILED DESCRIPTION:
Randomization will be performed using an external Interactive Web Response System. Subjects will be randomly assigned (1:1) in permuted blocks of different sizes, to have either BAX (Control group) or WALANT (Interventional group). A stratification of the randomization will be planned according to the Sex.

In the BAX group (usual technique), axillary brachial plexus block will be performed. In the WALANT group (experimental technique), local anesthesia will be performed. The Peripheral nerve blocks (PNBs) will be performed by a physician not involved in the peri-operative assessment. Care providers and outcomes assessors will be blinded to group allocation.

After obtaining venous access and placement of standard monitors, patients will be administered oxygen 2 L/min via nasal prongs. Thirty minutes before surgery, an experienced anesthesiologist will perform the regional blocks guided by ultrasound (Sonosite Export, Bothell, USA) using an ultrasound needle (Ultraplex 360°, B Braun, Melsungen, Germany) as follow:

* In the BAX group, patients will be placed in a supine position with their arm abducted to 90°. The ultrasound probe will be placed to obtain a transverse image of the axillary artery at the level of the conjoint tendon of the latissimus dorsi and teres major muscles. With an in-plane technique, a 50mm ultrasound needle (Ultraplex 360°, B Braun, Melsungen, Germany) will be advanced to achieve a spread of lidocaine (10mg/ml) around the musculocutaneous, radial, median and ulnar nerves. 30 ml of the solution will be used to achieve the BAX.
* In the WALANT group, patients will be placed in a supine position. Solution for local anesthesia will be prepared using 20 ml of lidocaine (10mg/ml) with epinephrine (0.005 mg/ml), 17 ml of saline solution and 3 ml of 8.4% sodium bicarbonate. The ultrasound probe will be placed to obtain a transverse image of the median nerve at the wrist. With an in-plane technique, a 50mm ultrasound needle (Ultraplex 360°, B Braun, Melsungen, Germany) will be advanced to achieve a spread of 5 ml of the solution posterior and then anterior to the median nerve under the annular carpal ligament. Then the ultrasound probe will be placed to obtain a longitudinal image of the median nerve at the wrist. With an in-plane technique, a 50mm ultrasound needle (Ultraplex 360°, B Braun, Melsungen, Germany) will be advanced to achieve a spread of 15 ml of the solution anterior to the median nerve towards the carpal tunnel. At last, a local infiltration with 5 ml of the solution will be performed around the surgical incision.

Upon completion of the blocks, patients will be transferred to the operating room.

In the operating room, a pneumatic tourniquet will be placed on the upper arm in all patients and will be inflated in patients of "BAX" group only. In case of pain or discomfort, an anesthetist blinded to treatment arm will decide on the need for an alternative anesthetic technique.

In ward:

* Postoperative analgesia protocol: systematic per os analgesia with paracetamol (1 g, 4 times a day) and ibuprofen (400 mg, 3 times a day)
* Mobilization of patient

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing endoscopic carpal tunnel release
* Consent for participation
* Affiliation to a social security system

Exclusion Criteria:

* Contraindication for regional anesthesia (truncal neuropathy, infection at the puncture site, coagulation disorder, …)
* Contraindication to any drugs used in the protocol (paracetamol, ketoprofen, propofol, lidocaine, epinephrine)
* Chronic pain syndrome
* Preoperative Anxiety
* Pregnant or breastfeeding women
* Patients under protection of the adults (guardianship, curators or safeguard of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
Regional anesthesia success | 2 hours
  Need (or not) for additional anesthetic procedure during surgery: analgesics, sedation, general anesthesia, local anesthetics

SECONDARY OUTCOMES:
Surgery duration | 2 hours
  Time (in minutes) between the skin incision and the wound dressing procedure.
Length of hospital stay | 24 hours
  Time (in minutes) between ward admission and discharge.
Discharge criteria assessed by PADSS | 24 hours
  Time (in minutes) between the regional anesthesia and the ability to discharge defined by the modified Post Anesthesia Discharge Scoring System (PADSS) who achieve a score of 9 or more.
Patient satisfaction assessed by EVAN-LR self-reported questionnaire | 24 hours
  EVAN-LR self-reported questionnaire comprising 19 items structured in five dimensions, depending on their content: Attention (4 items), Information (5 items), Discomfort (4 items), Waiting (2 items), and Pain (4 items). Each item is linearly transformed to a 0-100 scale, with 100 indicating the best possible level of satisfaction and 0 the worst.
Postoperative pain at the surgical site assessed by VRS | 24 hours
  Maximum postoperative pain at the surgical site will be assessed at Day-0 et at Day-1 using a Verbal Rating Scale (VRS) ranging from 0 to 10 (0=no pain, 10=worst possible pain).
Surgical site bleeding | 2 hours
  Surgeon's clear-field satisfactory score: 1=bloodless, 2=little blood, 3=bloody field but performable, 4=bloody field
Rate of complications | 24 hours
  Incidence of complications related to RA procedure: vascular puncture, paresthesia, local anesthetic systemic toxicity

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Médipôle Garonne, Toulouse, Haute-Garonne, France

REFERENCES:
- [Derived] Virtos M, Chassery C, Marty P, Basset B, Casalprim J, Vuillaume C, De Lussy A, Atthar V, Naudin C, Joshi G, Rontes O. Wide awake local anesthesia no tourniquet (WALANT) versus ultrasound-guided axillary block in carpal tunnel release: a non-inferiority randomized controlled trial. Reg Anesth Pain Med. 2025 Nov 13:rapm-2025-107152. doi: 10.1136/rapm-2025-107152. Online ahead of print. PMID 41233154